CLINICAL TRIAL: NCT03620292
Title: Cholangiocarcinoma Detection Using an Intraoperative Fluorescence Image Guided Approach With Bevacizumab-IRDye 800CW
Brief Title: Fluorescence Image Guided Surgery in Cholangiocarcinoma
Acronym: COUGAR
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, dr. W.B. Nagengast, MD, Dr. W.B. Nagengast, Gastroenterologist, Principal Investigator, University Medical Center Groningen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL65378.042.18
Record Dates: First submitted 2018-06-11; First posted 2018-08-08 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Hilar Cholangiocarcinoma
MeSH Terms: conditions — Klatskin Tumor | interventions — Optical Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intraoperative NIR fluorescence imaging (Experimental): A non-randomized, non-blinded, prospective, single center pilot dose escalation study with bevacizumab-800CW for NIR fluorescence image guided surgery in hilar cholangiocarcinoma
  * IV-administration of 10, 25 or 50 mg of the fluorescent tracer bevacizumab-800CW to a total of 15 patients with resectable hilar cholangiocarcinoma 3 days prior to surgery.
  * Peroperative open air NIR fluorescence imaging
  * Ex vivo endoscopic and histopathological NIR fluorescence imaging
  Interventions: Drug: Bevacizumab-IRDye800CW; Device: near infrared (NIR) fluorescence imaging

INTERVENTIONS:
Drug: Bevacizumab-IRDye800CW — Intravenous administration of Bevacizumab-IRDye800CW prior to surgery for hilar cholangiocarcinoma
  Other Names: Tracer administration
Device: near infrared (NIR) fluorescence imaging — Intraoperative NIR fluorescence imaging of hilar cholangiocarcinoma, lymph nodes, resection margins, resection specimens
  Other Names: optical imaging

SUMMARY:
Cholangiocarcinoma is an epithelial cell malignancy arising from varying locations within the biliary tree and is difficult to diagnose due to the often-silent clinical nature. The best chance of long-term survival and potential cure is surgical resection with negative surgical margins, but many patients are unresectable due to locally advanced or metastatic disease at diagnosis. Because cholangiocarcinoma is difficult to diagnose at an early stage and extends diffusely, most patients have unresectable disease at clinical presentation, and prognosis is very poor (5-year survival is 0-40% even in resected cases)

There is a need for better visualization of tumor tissue, lymph nodes and resection margins during surgery for perihilar cholangiocarcinoma (PHCC). Optical molecular imaging of PHCC associated biomarkers is a promising technique to accommodate this need. The biomarkers Vascular Endothelial Growth Factor (VEGF-A), Epidermal Growth Factor Receptor (EGFR) and c-MET are all overexpressed in PHCC versus normal tissue and are proven to be valid targets for molecular imaging. Currently, tracers that target these biomarkers are available for use in clinical studies. In previous studies with other tumor types, the investigators tested the tracer bevacizumab-IRDye800CW for the biomarker VEGF-A with very promising results. Since all markers show roughly similar expression in ex vivo studies, the initial study will be performed with bevacizumab-IRDye800CW as the investigators have the most experience with this tracer. The investigators hypothesize that the tracer bevacizumab-IRDye 800CW accumulates in PHCC tissue, enabling visualization using a NIR intraoperative camera system and ex vivo NIR endoscopy. In this pilot study, the investigators will determine if it is possible to detect PHCC intraoperatively and by ex vivo NIR endoscopy using bevacizumab 800CW, and which tracer dose gives the best target-to-background ratio. The most optimal tracer dose will be selected for a future phase II trial.

DETAILED DESCRIPTION:
See brief summary

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical suspicion of PHCC who are scheduled to undergo surgical intervention with curative intent
* WHO performance score 0-2.

Exclusion Criteria:

* Medical or psychiatric conditions that compromise the patient's ability to give informed consent.
* Other invasive malignancy
* Pregnant or lactating women.
* History of infusion reactions to bevacizumab or other monoclonal antibody therapies.
* Inadequately controlled hypertension with or without current antihypertensive medications
* Within 6 months prior to inclusion: myocardial infarction, TIA, CVA pulmonary embolism, uncontrolled chronic hepatic failure, unstable angina pectoris.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Optimal dose finding of Bevacizumab 800CW in hilar cholangiocarcinoma | 24 months
  - Comparison of three doses of Bevacizumab 800CW by calculating target to background ratios in fluorescence images obtained during and directly after the surgical procedure and fluorescence images obtained during ex vivo analyses in bread loaf slices and in histological slices (odyssey scanner, fluorescence microscopy).

SECONDARY OUTCOMES:
Peroperative detection of hilar cholangiocarcinoma with real-time near-infrared fluorescence camera | 24 months
  - Comparison between perioperative fluorescent imaging and ex vivo analysis (histology, breadloaf slices) to see if detection of tumor tissue is feasible. I.e. is high fluorescent signal corresponding with localization of tumor tissue in ex-vivo analysis?
Detection of hilar cholangiocarcinoma in real-time near-infrared fluorescence ex-vivo endoscopy | 24 months
  - Comparison of endoscopic fluorescent imaging and ex vivo analysis(histology, breadloaf slices) to see if endoscopic detection is feasible. I.e. is high fluorescent signal seen during ex-vivo endoscopy corresponding with localization of tumor tissue in ex-vivo analysis?
Establish tracer distribution in tumour tissue | 24 months
  - Visualisation of tracer distribution at microscopic level using ex vivo needle based confocal laser endomicroscopy.
Measurement of fluorescence in tumour tissue en surrounding normal tissue | 24 months
  - Correction for scattering and measurement of fluorescent signal using spectroscopy ex vivo.

CONTACTS AND LOCATIONS:
Overall Officials: G. M. van Dam, MD, PhD, Principal Investigator — University Medical Center Groningen; M. T. de Boer, MD, PhD, Principal Investigator — University Medical Center Groningen; W. B. Nagengast, MD, PhD, PharmD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No